CLINICAL TRIAL: NCT02277600
Title: Open-Label, Single-Sequence, Two-Cohort Study to Evaluate the Effect of Darunavir/Cobicistat and Cobicistat on BMS-626529 in Healthy Subjects
Brief Title: A Phase 1 Antiretroviral Drug-Drug Interaction Study in Healthy Volunteers (DDI)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 206285; AI438-044 (Other: Bristol-Myers Squibb)
Record Dates: First submitted 2014-10-27; First posted 2014-10-29 (Estimated); Last update posted 2018-01-24 (Actual); Status verified 2017-07

CONDITIONS: Infection, Human Immunodeficiency Virus
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome | interventions — fostemsavir; Darunavir; Cobicistat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1, Treatment A, B (Experimental): Treatment A:
  BMS-663068 orally twice daily (BID) on Days 1 through 4
  Treatment B:
  BMS-663068 orally BID plus DRV/COBI orally once daily (QD) on Days 5 through 14
  Interventions: Drug: BMS-663068; Drug: Darunavir; Drug: Cobicistat
- Cohort 2, Treatment C, D (Experimental): Treatment C:
  BMS-663068 orally BID on Days 1 through 4
  Treatment D:
  BMS-663068 orally BID plus COBI QD on Days 5 through 14
  Interventions: Drug: BMS-663068; Drug: Cobicistat

INTERVENTIONS:
Drug: BMS-663068 — BMS-663068
Drug: Darunavir — Darunavir
  Arms: Cohort 1, Treatment A, B
Drug: Cobicistat — Cobicistat

SUMMARY:
This is an open-label, single sequence, 2-cohort, drug-drug interaction study in healthy male and female subjects. There is no formal hypothesis, however, it is expected that the coadministration of BMS-663068 with darunavir (DRV)/cobicistat (COBI) or COBI will increase the systemic exposure of BMS-626529.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female
* Nonsmoking subjects
* Ages 18 to 50 years
* Inclusive with a body mass index of 18.0 to 32.0 kg/m2, inclusive
* Women of childbearing potential
* Must agree to follow instructions for methods of contraception for the duration of the study plus 34 days post-treatment completion

Exclusion Criteria:

* Any history of acute or chronic medical and surgical illness.
* Personal of family history of hemophilia A or B
* Other protocol defined exclusion criteria could apply

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2014-11-05 (Actual); Primary Completion 2015-01-12 (Actual); Study Completion 2015-01-12 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters (maximum observed plasma concentration and area under the concentration-time curve in 1 dosing interval) for BMS-626529 | predose and up to 12 hours post dose on Days 4 and 14
  In the presence or absence of multiple doses of DRV/COBI or COBI

OTHER OUTCOMES:
Safety as assessed by adverse events and other physical parameters | From dosing (Day 1) to Day 14
  Collection of adverse events and other physical parameters to assess safety and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (1):
- GSK Investigational Site, San Antonio, Texas, United States

REFERENCES:
- [Derived] Moore K, Thakkar N, Magee M, Sevinsky H, Vakkalagadda B, Lubin S, Llamoso C, Ackerman P. Pharmacokinetics of Temsavir, the Active Moiety of the HIV-1 Attachment Inhibitor Prodrug, Fostemsavir, Coadministered with Cobicistat, Etravirine, Darunavir/Cobicistat, or Darunavir/Ritonavir with or without Etravirine in Healthy Participants. Antimicrob Agents Chemother. 2022 Apr 19;66(4):e0225121. doi: 10.1128/aac.02251-21. Epub 2022 Mar 22. PMID 35315687